CLINICAL TRIAL: NCT05106257
Title: Optimizing Self-management COPD Treatment Through the American Lung Association Helpline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20050506
Record Dates: First submitted 2021-10-12; First posted 2021-11-03 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Copd
Keywords: COPD; Self-management; Lifestyle change; Patient education; Quality of life; Physical activity; Inhaler use; Caregiver support
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition #1 (Experimental): Education = short Walking training = on Inhaler training = on Caregiver support = on
  Interventions: Behavioral: Self-management education (short); Behavioral: Ground-based walking training; Behavioral: Inhaler training; Behavioral: Caregiver support
- Condition #2 (Experimental): Education = short Walking training = on Inhaler training = on Caregiver support = off
  Interventions: Behavioral: Self-management education (short); Behavioral: Ground-based walking training; Behavioral: Inhaler training
- Condition #3 (Experimental): Education = short Walking training = on Inhaler training = off Caregiver support = on
  Interventions: Behavioral: Self-management education (short); Behavioral: Ground-based walking training; Behavioral: Caregiver support
- Condition #4 (Experimental): Education = short Walking training = on Inhaler training = off Caregiver support = off
  Interventions: Behavioral: Self-management education (short); Behavioral: Ground-based walking training
- Condition #5 (Experimental): Education = short Walking training = off Inhaler training = on Caregiver support = on
  Interventions: Behavioral: Self-management education (short); Behavioral: Inhaler training; Behavioral: Caregiver support
- Condition #6 (Experimental): Education = short Walking training = off Inhaler training = on Caregiver support = off
  Interventions: Behavioral: Self-management education (short); Behavioral: Inhaler training
- Condition #7 (Experimental): Education = short Walking training = off Inhaler training = off Caregiver support = on
  Interventions: Behavioral: Self-management education (short); Behavioral: Caregiver support
- Condition #8 (Experimental): Education = short Walking training = off Inhaler training = off Caregiver support = off
  Interventions: Behavioral: Self-management education (short)
- Condition #9 (Experimental): Education = long Walking training = on Inhaler training = on Caregiver support = on
  Interventions: Behavioral: Ground-based walking training; Behavioral: Inhaler training; Behavioral: Caregiver support; Behavioral: Self-management education (long)
- Condition #10 (Experimental): Education = long Walking training = on Inhaler training = on Caregiver support = off
  Interventions: Behavioral: Ground-based walking training; Behavioral: Inhaler training; Behavioral: Self-management education (long)
- Condition #11 (Experimental): Education = long Walking training = on Inhaler training = off Caregiver support = on
  Interventions: Behavioral: Ground-based walking training; Behavioral: Caregiver support; Behavioral: Self-management education (long)
- Condition #12 (Experimental): Education = long Walking training = on Inhaler training = off Caregiver support = off
  Interventions: Behavioral: Ground-based walking training; Behavioral: Self-management education (long)
- Condition #13 (Experimental): Education = long Walking training = off Inhaler training = on Caregiver support = on
  Interventions: Behavioral: Inhaler training; Behavioral: Caregiver support; Behavioral: Self-management education (long)
- Condition #14 (Experimental): Education = long Walking training = off Inhaler training = on Caregiver support = off
  Interventions: Behavioral: Inhaler training; Behavioral: Self-management education (long)
- Condition #15 (Experimental): Education = long Walking training = off Inhaler training = off Caregiver support = on
  Interventions: Behavioral: Caregiver support; Behavioral: Self-management education (long)
- Condition #16 (Experimental): Education = long Walking training = off Inhaler training = off Caregiver support = off
  Interventions: Behavioral: Self-management education (long)

INTERVENTIONS:
Behavioral: Self-management education (short) — The self-management education condition is based on the Living Well with COPD program. The program consists of a mailed booklet and structured phone counseling delivered by certified COPD educators. Topics include disease information, breathing retraining, action planning, medication use, energy conservation, and following good health habits. The short condition consists of two calls (30-45 minutes each) to introduce patient education topics and refer to the booklet for further information.
  Arms: Condition #1; Condition #2; Condition #3; Condition #4; Condition #5; Condition #6; Condition #7; Condition #8
Behavioral: Ground-based walking training — Participants randomized to this condition will be mailed a pedometer (3DFitBud Simple Step Counter) and instructed on its use to establish baseline steps/ day for 7 days. They will then receive a booklet with instructions to establish a walking program and three brief (10-15 minute), bi-weekly calls from a trained staff member to review step count values and engage in setting personal activity goals over the course of 6 weeks, following established exercise guidelines for individuals with COPD.
  Arms: Condition #1; Condition #10; Condition #11; Condition #12; Condition #2; Condition #3; Condition #4; Condition #9
Behavioral: Inhaler training — Participants randomized to this condition will receive two sessions of inhaler technique education using a virtual teach-to-goal (TTG) method in which individuals are observed using their inhaler, provided feedback, and then observed again.
  Arms: Condition #1; Condition #10; Condition #13; Condition #14; Condition #2; Condition #5; Condition #6; Condition #9
Behavioral: Caregiver support — Participants randomized to this condition will identify an informal caregiver who is involved in their healthcare (i.e., spouse, family member, or friend), who will receive a mailed copy of the Respiratory Health Association's COPD Caregiver's Toolkit, a comprehensive informational resource to support the care of the person living with COPD. Caregivers will receive two brief (10-15 minute) check-in calls from a trained staff member. The structured content of these sessions will include providing an overview of toolkit content, identifying goals for sections(s) to review and incorporate into caregiving activities, and addressing any questions.
  Arms: Condition #1; Condition #11; Condition #13; Condition #15; Condition #3; Condition #5; Condition #7; Condition #9
Behavioral: Self-management education (long) — The self-management education condition is based on the Living Well with COPD program. The program consists of a mailed booklet and structured phone counseling delivered by certified COPD educators. Topics include disease information, breathing retraining, action planning, medication use, energy conservation, and following good health habits. The long condition consists of five, weekly calls (30-45 minutes each) following a structured curriculum of patient education topics.
  Arms: Condition #10; Condition #11; Condition #12; Condition #13; Condition #14; Condition #15; Condition #16; Condition #9

SUMMARY:
Although self-management treatment improves quality of life among individuals with COPD, there is limited understanding of which elements of treatment are most effective. The proposed research will test the feasibility of using an engineering-inspired study design to identify effective COPD self-management treatment components. The long-term goal of this line of research is to optimize the effectiveness of COPD self-management treatment, and improve quality of life for individuals with COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is an increasingly prevalent and costly chronic health condition, and is the third major cause of morbidity and mortality in the United States. Self-management treatment programs for COPD are shown to improve health-related quality of life and prevent COPD-related hospitalizations. Despite their clinical benefits, these programs are typically multi-component and time- and resource-intensive. To date, no study has been conducted to isolate the role of individual self-management treatment components in contributing to improved COPD outcomes. The proposed research will establish the feasibility of using the Multiphase Optimization Strategy (MOST) framework to optimize COPD self-management treatment delivered by the American Lung Association (ALA) Helpline. Treatment components to be evaluated include duration of self-management education, ground-based walking training, inhaler training, and caregiver support. The primary outcome is health-related quality of life, with secondary outcomes of COPD symptom burden, self-management behaviors, and hospitalization. Specific aims are:

Aim 1: Design a factorial experiment and develop operational procedures. The investigators will design a factorial experiment with the same number of experimental conditions and length of follow-up as the planned optimization trial. In collaboration with the ALA COPD Helpline, the investigators will develop operational procedures (i.e., recruitment, screening, randomization, and database management) for successful implementation.

Aim 2: Establish feasibility and acceptability by pilot testing the study design. The investigators will deliver treatment to three participants per experimental condition (N=48) with good fidelity, and will remotely assess baseline, mediator, and outcome variables. The investigators will conduct qualitative interviews at end-of-treatment with 15-20 participants. Resulting values will provide estimates of recruitment and retention rates, treatment fidelity, acceptability of treatment components, and outcome measure variability to inform a subsequent, fully-powered optimization trial. The primary outcome is health-related quality of life, with secondary outcomes of COPD symptom burden, self-management behaviors, and hospitalization.

ELIGIBILITY:
Inclusion criteria:

Eligible participants will be males and females who are:

1. 40 years or older,
2. report a physician diagnosis of COPD,
3. use an inhaler for COPD at least once a week,
4. able to walk at least one block without assistance,
5. able to identify a caregiver, and
6. have access to a connected device (i.e., smart phone, tablet, and/ or computer).

Exclusion criteria:

1. cognitive dysfunction impairing ability to provide informed consent and follow study procedures,
2. terminal illness (i.e. less than 6 months life expectancy) that is non-COPD related,
3. living at a chronic care facility (i.e. nursing home, assisted living), or
4. inability to speak and read English.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda R Mathew, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Condition #1: Education = short Walking training = on Inhaler training = on Caregiver support = on
  Self-management education (short): The self-management education condition is based on the Living Well with COPD program. The program consists of a mailed booklet and structured phone counseling delivered by certified COPD educators. The short condition consists of two calls (30-45 minutes each).
  Ground-based walking training: Participants randomized to this condition will be mailed a pedometer and instructed on its use to establish baseline steps/ day for 7 days. They will then receive a booklet with instructions to establish a walking program and three brief (10-15 minute), bi-weekly calls from a trained staff member to review step count values and engage in setting personal activity goals over the course of 6 weeks.
  Inhaler training: Participants randomized to this condition will receive two sessions of inhaler technique education using a virtual teach-to-goal (TTG) method in which individuals are observed using their inhaler, provided feedback, and then observed again.
  Caregiver support: Participants randomized to this condition will identify an informal caregiver (i.e., spouse, family member, or friend), who will receive a mailed copy of the Respiratory Health Association's COPD Caregiver's Toolkit. Caregivers will receive two brief (10-15 minute) check-in calls from a trained staff member.
- Condition #3: Education = short Walking training = on Inhaler training = off Caregiver support = on
  Self-management education (short): The self-management education condition is based on the Living Well with COPD program. The program consists of a mailed booklet and structured phone counseling delivered by certified COPD educators. The short condition consists of two calls (30-45 minutes each).
  Ground-based walking training: Participants randomized to this condition will be mailed a pedometer and instructed on its use to establish baseline steps/ day for 7 days. They will then receive a booklet with instructions to establish a walking program and three brief (10-15 minute), bi-weekly calls from a trained staff member to review step count values and engage in setting personal activity goals over the course of 6 weeks.
  Caregiver support: Participants randomized to this condition will identify an informal caregiver (i.e., spouse, family member, or friend), who will receive a mailed copy of the Respiratory Health Association's COPD Caregiver's Toolkit. Caregivers will receive two brief (10-15 minute) check-in calls from a trained staff member.
- Condition #5: Education = short Walking training = off Inhaler training = on Caregiver support = on
  Self-management education (short): The self-management education condition is based on the Living Well with COPD program. The program consists of a mailed booklet and structured phone counseling delivered by certified COPD educators. The short condition consists of two calls (30-45 minutes each).
  Inhaler training: Participants randomized to this condition will receive two sessions of inhaler technique education using a virtual teach-to-goal (TTG) method in which individuals are observed using their inhaler, provided feedback, and then observed again.
  Caregiver support: Participants randomized to this condition will identify an informal caregiver (i.e., spouse, family member, or friend), who will receive a mailed copy of the Respiratory Health Association's COPD Caregiver's Toolkit. Caregivers will receive two brief (10-15 minute) check-in calls from a trained staff member.
- Condition #9: Education = long Walking training = on Inhaler training = on Caregiver support = on
  Ground-based walking training: Participants randomized to this condition will be mailed a pedometer and instructed on its use to establish baseline steps/ day for 7 days. They will then receive a booklet with instructions to establish a walking program and three brief (10-15 minute), bi-weekly calls from a trained staff member to review step count values and engage in setting personal activity goals over the course of 6 weeks.
  Inhaler training: Participants randomized to this condition will receive two sessions of inhaler technique education using a virtual teach-to-goal (TTG) method in which individuals are observed using their inhaler, provided feedback, and then observed again.
  Caregiver support: Participants randomized to this condition will identify an informal caregiver (i.e., spouse, family member, or friend), who will receive a mailed copy of the Respiratory Health Association's COPD Caregiver's Toolkit. Caregivers will receive two brief (10-15 minute) check-in calls from a trained staff member.
  Self-management education (long): The self-management education condition is based on the Living Well with COPD program. The program consists of a mailed booklet and structured phone counseling delivered by certified COPD educators. The long condition consists of five, weekly calls (30-45 minutes each).
- Condition #11: Education = long Walking training = on Inhaler training = off Caregiver support = on
  Ground-based walking training: Participants randomized to this condition will be mailed a pedometer and instructed on its use to establish baseline steps/ day for 7 days. They will then receive a booklet with instructions to establish a walking program and three brief (10-15 minute), bi-weekly calls from a trained staff member to review step count values and engage in setting personal activity goals over the course of 6 weeks.
  Caregiver support: Participants randomized to this condition will identify an informal caregiver (i.e., spouse, family member, or friend), who will receive a mailed copy of the Respiratory Health Association's COPD Caregiver's Toolkit. Caregivers will receive two brief (10-15 minute) check-in calls from a trained staff member.
  Self-management education (long): The self-management education condition is based on the Living Well with COPD program. The program consists of a mailed booklet and structured phone counseling delivered by certified COPD educators. The long condition consists of five, weekly calls (30-45 minutes each).
- Condition #13: Education = long Walking training = off Inhaler training = on Caregiver support = on
  Inhaler training: Participants randomized to this condition will receive two sessions of inhaler technique education using a virtual teach-to-goal (TTG) method in which individuals are observed using their inhaler, provided feedback, and then observed again.
  Caregiver support: Participants randomized to this condition will identify an informal caregiver (i.e., spouse, family member, or friend), who will receive a mailed copy of the Respiratory Health Association's COPD Caregiver's Toolkit. Caregivers will receive two brief (10-15 minute) check-in calls from a trained staff member.
  Self-management education (long): The self-management education condition is based on the Living Well with COPD program. The program consists of a mailed booklet and structured phone counseling delivered by certified COPD educators. The long condition consists of five, weekly calls (30-45 minutes each).
Period: Overall Study
Arm/Group | Condition #1 | Condition #2 | Condition #3 | Condition #4 | Condition #5 | Condition #6 | Condition #7 | Condition #8 | Condition #9 | Condition #10 | Condition #11 | Condition #12 | Condition #13 | Condition #14 | Condition #15 | Condition #16
Started | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition #1 | Condition #2 | Condition #3 | Condition #4 | Condition #5 | Condition #6 | Condition #7 | Condition #8 | Condition #9 | Condition #10 | Condition #11 | Condition #12 | Condition #13 | Condition #14 | Condition #15 | Condition #16 | Total
Number analyzed (Participants) | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (13) | 58 (11) | 63 (2) | 66 (7) | 67 (11) | 67 (1) | 65 (8) | 65 (5) | 61 (27) | 63 (14) | 70 (9) | 64 (8) | 74 (4) | 71 (9) | 74 (1) | 74 (7) | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 1 | 2 | 28
  Male | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 2 | 1 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 3 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 13
  White | 2 | 1 | 0 | 2 | 2 | 3 | 1 | 3 | 1 | 2 | 3 | 2 | 3 | 2 | 0 | 3 | 30
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 46

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life
Description: Measured by the Chronic Respiratory Disease Questionnaire (CRQ) dyspnea subscale score. Possible scale range is 1-7; higher scores indicate better health-related quality of life.
Time Frame: Change from baseline at 90-day follow-up
Population: Please note that the Arms/ Groups in the Outcome Measures are a recombination of the Participant Flow Arms/ Groups to report results by factor.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ground-based Walking Training (on): Ground-based walking training: Participants randomized to this condition will be mailed a pedometer (3DFitBud Simple Step Counter) and instructed on its use to establish baseline steps/ day for 7 days. They will then receive a booklet with instructions to establish a walking program and three brief (10-15 minute), bi-weekly calls from a trained staff member to review step count values and engage in setting personal activity goals over the course of 6 weeks, following established exercise guidelines for individuals with COPD.
- Ground-based Walking Training (Off): Not randomized to receive ground-based walking training.
- Inhaler Training (on): Inhaler training: Participants randomized to this condition will receive two sessions of inhaler technique education using a virtual teach-to-goal (TTG) method in which individuals are observed using their inhaler, provided feedback, and then observed again.
- Inhaler Training (Off): Not randomized to receive inhaler training
- Caregiver Support (on): Caregiver support: Participants randomized to this condition will identify an informal caregiver (i.e., spouse, family member, or friend), who will receive a mailed copy of the Respiratory Health Association's COPD Caregiver's Toolkit. Caregivers will receive two brief (10-15 minute) check-in calls from a trained staff member.
- Caregiver Support (Off): Not randomized to receive caregiver support
Arm/Group | Self-management Education (Short) | Self-management Education (Long) | Ground-based Walking Training (on) | Ground-based Walking Training (Off) | Inhaler Training (on) | Inhaler Training (Off) | Caregiver Support (on) | Caregiver Support (Off)
Number analyzed (Participants) | 22 | 24 | 22 | 24 | 23 | 23 | 23 | 23
score on a scale | 0.6 (1.5) | 0.7 (1.5) | 1.3 (1.5) | 0.1 (1.2) | 0.3 (1.6) | 0.9 (1.3) | 0.7 (1.5) | 0.5 (1.4)

2. Secondary Outcome: COPD Symptom Burden
Description: Measured by the COPD Assessment Test (CAT), an 8-item questionnaire measuring the global impact of dyspnea on health status. Possible score range is 0-40; higher scores indicate more severe symptom impact.
Time Frame: Change from baseline at 90-day follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-management Education (Short) | Self-management Education (Long) | Ground-based Walking Training (on) | Ground-based Walking Training (Off) | Inhaler Training (on) | Inhaler Training (Off) | Caregiver Support (on) | Caregiver Support (Off)
Number analyzed (Participants) | 19 | 18 | 15 | 22 | 17 | 20 | 19 | 18
units on a scale | -1.9 (6) | -3.1 (5) | -3.9 (4.9) | -1.5 (5.8) | -0.4 (4.3) | -4.3 (5.9) | -0.6 (4.5) | -4.4 (5.9)

3. Secondary Outcome: Self-management Behaviors
Description: Measured by the Patient Activation Measure (PAM-13), a 13-item questionnaire measuring patient knowledge, skill, and confidence for self-management. Items are summed to yield a raw score (possible range 13-52), which is then converted to a normalized score (possible range 0-100). Higher scores indicate better self-management.
Time Frame: Change from baseline at 90-day follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-management Education (Short) | Self-management Education (Long) | Ground-based Walking Training (on) | Ground-based Walking Training (Off) | Inhaler Training (on) | Inhaler Training (Off) | Caregiver Support (on) | Caregiver Support (Off)
Number analyzed (Participants) | 16 | 16 | 13 | 19 | 13 | 19 | 16 | 16
score on a scale | 3.6 (18) | 12.7 (16.9) | 10.9 (17.9) | 6.2 (18) | 3.1 (20.9) | 11.6 (15) | 8.3 (13.9) | 8 (21.5)

4. Secondary Outcome: Hospitalization
Description: Self-reported hospitalization history.
Time Frame: Incidence at 90-day follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Self-management Education (Short) | Self-management Education (Long) | Ground-based Walking Training (on) | Ground-based Walking Training (Off) | Inhaler Training (on) | Inhaler Training (Off) | Caregiver Support (on) | Caregiver Support (Off)
Number analyzed (Participants) | 22 | 24 | 22 | 24 | 23 | 23 | 23 | 23
Participants | 2 | 2 | 3 | 1 | 4 | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Self-management Education (Short) | Self-management Education (Long) | Ground-based Walking Training (on) | Ground-based Walking Training (Off) | Inhaler Training (on) | Inhaler Training (Off) | Caregiver Support (on) | Caregiver Support (Off)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24 | 0/22 | 0/24 | 0/23 | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 6/22 | 2/24 | 7/22 | 1/24 | 6/23 | 2/23 | 2/23 | 6/23
Other Adverse Events (participants affected / at risk) | 6/22 | 10/24 | 9/22 | 7/24 | 6/23 | 10/23 | 7/23 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-management Education (Short) (N=22) | Self-management Education (Long) (N=24) | Ground-based Walking Training (on) (N=22) | Ground-based Walking Training (Off) (N=24) | Inhaler Training (on) (N=23) | Inhaler Training (Off) (N=23) | Caregiver Support (on) (N=23) | Caregiver Support (Off) (N=23)
COPD exacerbation/ hospitalization (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 7 (7) | 1 (1) | 6 (6) | 2 (2) | 2 (2) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-management Education (Short) (N=22) | Self-management Education (Long) (N=24) | Ground-based Walking Training (on) (N=22) | Ground-based Walking Training (Off) (N=24) | Inhaler Training (on) (N=23) | Inhaler Training (Off) (N=23) | Caregiver Support (on) (N=23) | Caregiver Support (Off) (N=23)
Symptoms requiring immediate medical attention (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10) | 9 (9) | 7 (7) | 6 (6) | 10 (10) | 7 (7) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT05106257/Prot_SAP_000.pdf